CLINICAL TRIAL: NCT00160004
Title: The Effect of Intensive Controlled Exercise in the Early Stages of Amyotrophic Lateral Sclerosis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: problems with including patients and a large multicenter Trial is now starting as follow-up
Sponsor: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALSICEJ1
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2009-06-08 (Estimated); Status verified 2009-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Exercise; Fatigue; Quality-of-life
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Activity; Fatigue

INTERVENTIONS:
Behavioral: Intensive Controlled Exercise

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is a progressive neurological disorder characterized by amongst others asymmetric muscle weakness, respiratory insufficiency and spasticity. The disease is usually fatal within 2-3 years and until now there is no cure. ALS patients are usually supported by a multidisciplinary team. One of the members of this team is the physical therapist. The aim of physical therapy might be to enhance or to preserve cardiovascular fitness and muscle strength. Some authors suggest, however, that a moderate to high intensive exercise programme might lead to overuse weakness (an undesired fast progression of muscle weakness). The primary objective of this study is therefore to investigate whether regular moderate to high intensity exercise program in ALS can maintain or optimize cardiorespiratory fitness and muscle strength. A secondary objective is to investigate whether such a programme leads to overuse weakness and if there is a positive influence on patient's disability, fatigue and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Older dan 18 years Written Informed Consent Don't use walking adds such as a cane Patients must met El Escorial criteria for probable or definite ALS

Exclusion Criteria:

* Patients who are depending on intermittent or continuous mechanical ventilation Patients who are not able to understand and conform to the instructions Patients who already perform an exercise programme that can compare with our study Patients who have severe cardiopulmonary problems, DM or other problems concerning connective tissue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-03; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness measured with Astrand submaximal test

SECONDARY OUTCOMES:
Muscle Strength measured with MVIC (Maximum Voluntary Isometric Contraction)
Functional status measured with ALS-FRS-r Rating scale
Quality of life with ALS-AQ40 Questionnaire
Fatigue measured with CIS Questionnaire
Pulmonary function measured with FVC

CONTACTS AND LOCATIONS:
Overall Officials: Marten Munneke, PhD, Principal Investigator — Institute of Neurology, Radboud University Nijmegen Medical Centre, The Netherlands
Locations (1):
- Department of Allied health Occupations, Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Drory VE, Goltsman E, Reznik JG, Mosek A, Korczyn AD. The value of muscle exercise in patients with amyotrophic lateral sclerosis. J Neurol Sci. 2001 Oct 15;191(1-2):133-7. doi: 10.1016/s0022-510x(01)00610-4. PMID 11677004